CLINICAL TRIAL: NCT03411629
Title: Significance of Collections Around Colon in Patients With Acute Necrotizing Pancreatitis: a Prospective Study
Brief Title: Significance of Collections Around Colon in Patients With Acute Necrotizing Pancreatitis
Status: Completed | Type: Observational
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Mohan Gurjar, Additional Professor, Sanjay Gandhi Postgraduate Institute of Medical Sciences
Other Study IDs: 2017-235-IP-EXP
Record Dates: First submitted 2018-01-13; First posted 2018-01-26 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Acute Necrotizing Pancreatitis
Keywords: Necrotizing Pancreatitis; Critically ill; Mortality
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute pancreatitis is an inflammatory process which causes a local and systemic inflammatory response syndrome (SIRS). Although the majority of patients have a mild disease course, around 20% will develop moderate or severe pancreatitis, with necrosis of the (peri) pancreatic tissue and/or multiple-organ failure. Previous studies have correlated colonic involvement as a prognostic marker in acute pancreatitis. It is well known that translocation of the colonic flora may significantly influence the clinical course of patients with acute pancreatitis. The correlation between collection(s) around colon in CT finding and clinical outcomes has not been studied in necrotizing pancreatitis. In current study, the investigators will do a prospective observational study correlating collection(s) around the colon and clinical course of patients in acute necrotizing pancreatitis.

DETAILED DESCRIPTION:
Introduction and rationale of the study:

Acute pancreatitis is the leading gastrointestinal cause of hospitalization in the US, with 270,000 admissions annually. Acute pancreatitis is an inflammatory process which causes a local and systemic inflammatory response syndrome (SIRS). Although the majority of patients have a mild disease course, around 20% will develop moderate or severe pancreatitis, with necrosis of the (peri) pancreatic tissue and/or multiple-organ failure About 5-10% of patients develop necrosis of the pancreatic parenchyma, the peripancreatic tissue or both. A collection containing variable amounts of both fluid and necrosis associated with necrotizing pancreatitis; the necrosis can involve the pancreatic parenchyma and/or the peri- pancreatic tissues. A mature, encapsulated collection of pancreatic and/or peri- pancreatic necrosis with well defined inflammatory wall is walled off necrosis (WON). It usually occurs >4 weeks after onset of necrotizing pancreatitis.

Colonic involvement may predict disease severity and outcome. Clinical features may appear late in the course. Colonic complications occur in 1% patients with acute pancreatitis with 6-40% occurring with necrotizing pancreatitis. Correlation between colonic wall thickening at CT and the clinical course has already been established in non-necrotizing pancreatitis. Colonic necrosis is an adverse prognostic factor in pancreatic necrosis. Extension of necrosis towards the transverse colon and the splenic flexure were seen most commonly observed.

Previous studies have correlated colonic involvement as a prognostic marker in acute pancreatitis. It is well known that translocation of the colonic flora may significantly influence the clinical course of patients with acute pancreatitis. The correlation between collection(s) around colon in CT finding and clinical outcomes has not been studied in necrotizing pancreatitis.

Work plan methodology:

This will be a prospective, observational study, to be conducted in 20 bed ICU of department of Critical Care Medicine, Sanjay Gandhi Institute of Postgraduate and Medical Sciences, Lucknow.

All adult (≥18 years) ICU patients who had acute necrotizing pancreatitis will be considered. Demographic and clinical characteristics of all ICU patients who fulfill inclusion criteria will be collected along with relevant laboratory tests done for patient management routinely. ICU prognostication scores, i.e., Acute Physiologic and Chronic Health Evaluation (APACHE) II score and Sequential Organ Failure Assessment (SOFA) score will also be recorded. The investigators will review all available computed tomography scans (CT Scans) of abdomen, from 2nd week to 6th week of pancreatitis, which will be done as per treating clinicians during patient ICU stay.

Collection around colon is classified as: 1. No pericolonic collection; 2. Less than 90 degree encasement of colon; 3. In between 90-180 degree; 4. More than 180 degree encasement of colon. Other intra-abdominal collection will also be noted along with mesocolon.

Clinical course will be followed till ICU discharge in terms of need for drain and surgery, intra-abdominal infection, and survival at discharge.

Statistical analysis: Descriptive analysis will be done and data will be presented as mean or median.

Intervention: None. Waiver of consent has been granted by the Institute Ethics Committee (IEC).

ELIGIBILITY:
Inclusion Criteria:

* All adult (≥18 years) ICU patients who had acute necrotizing pancreatitis will be considered.

Exclusion Criteria:

* Age <18 years
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult (≥18 years) ICU patients who had acute necrotizing pancreatitis.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-05-18 (Actual)

PRIMARY OUTCOMES:
Correlating collection(s) around the colon and clinical course of patients in acute necrotizing pancreatitis. | Up to 6 weeks of the acute pancreatitis
  To study CT finding of collection(s) around colon in patients with acute necrotizing pancreatitis and its association with clinical course i.e. intra-abdominal infection, need of drain/surgery and survival at ICU discharge..

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Gurjar, MD, PDCC, Principal Investigator — Sanjay Gandhi Postgraduate Institute of Medical Sciences (SGPGIMS)
Locations (1):
- Department of Critical Care Medicine, SGPGIMS, Lucknow, Uttar Pradesh, India